CLINICAL TRIAL: NCT02913677
Title: Prolonged Minimal Enteral Nutrition Versus Slowly Advancing Enteral Nutrition in Very Low Birth Weight Infants:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZTB7915
Record Dates: First submitted 2016-08-15; First posted 2016-09-26 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2016-08

CONDITIONS: Enteral Nutrition; Born Very Premature; Infant, Very Low Birth Weight
Keywords: feeding intolerance; minimal enteral nutrition; very low birth weight; preterm infant
MeSH Terms: conditions — Premature Birth | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Active Comparator): prolonged minimal enteral nutrition
  Interventions: Dietary Supplement: nutrition
- group 2 (Placebo Comparator): slowly advancing enteral nutrition
  Interventions: Dietary Supplement: nutrition

INTERVENTIONS:
Dietary Supplement: nutrition — Feeding was started in the first 48 hours. Fed with 10-15 ml/kg/d MEN for 5 days and than feed volumes were advanced by 20-25 ml/kg/d until 150ml/kg/d feed volume was achieved.

SUMMARY:
Recent studies showed the benefits of early initiation and advancement enteral feeds with daily increments in preterm infants on decreasing invasive infections and early achievement of full enteral feedings. But the data on enteral feeds of extremely low birthweight infants are limited. Preterm infants especially those <1250 gr birthweight are at increased risk of developing feeding intolerance and necrotizing enterocolitis (NEC) and so the initiation and the rate of increments of enteral feeds are usually uncertain issues for neonatologists.

DETAILED DESCRIPTION:
Background: Recent studies showed the benefits of early initiation and advancement enteral feeds with daily increments in preterm infants on decreasing invasive infections and early achievement of full enteral feedings. But the data on enteral feeds of extremely low birthweight infants are limited. Preterm infants especially those <1250 gr birthweight are at increased risk of developing feeding intolerance and necrotizing enterocolitis and so the initiation and the rate of increments of enteral feeds are usually uncertain issues for neonatologists.

Aim: To assess the effects of two different feeding strategies in very low birth weight preterm infants with birth weight ≤1250 gr and gestational age ≤32 weeks on the incidence of feeding intolerance and time to reach full enteral feedings.

Study design: prospective randomized controlled trial comparing the effects of prolonged minimal enteral nutrition (MEN) with progressive advancing enteral feedings.

Primary outcomes: incidence of feeding intolerance and time to reach full enteral feedings sustained for 72 hours.

Secondary outcomes: incidence of NEC, sepsis, duration of hospitalization Methods: a total of 200 preterm infants with gestational age ≤32 weeks and birthweight ≤1250 gr were randomly allocated to one of the 2 feeding strategies.

Group 1-) Feeding was started in the first 48 hours. Fed with 10-15 ml/kg/d MEN for 5 days and than feed volumes were advanced by 20-25 ml/kg/d until 150ml/kg/d feed volume was achieved.

Group 2-) Feeding was started in the first 48 hours with a volume of 10-15 ml/kg/d and advanced with daily increments of 20-25 ml/kg/d until 150 ml/kg/d feed volume was achieved.

MEN was withheld when the infant developped NEC or when there was bilious emesis or gross blood in stool.

Feeding intolerance was defined as; Bilious emesis or gastric residuals Grossly bloody stools, Abdominal tenderness or discoloration, Gastric residuals in ≥%50 of previous feed volume Emesis ≥3 times in 8 hours period Clinical or radiological evidence of NEC When feeding intolerance was developped feeds were withheld in both groups until the problem was resolved and resumed feed volume where withheld.

In the study unit parenteral nutrition was started on the first day of birth. Parenteral nutrition volume was decreased as the enteral feeds increased. Breast milk was the first choice for enteral nutrition if available but if not preterm formulas were used. When 100ml/kg/d enteral feed volume was achieved breast milk was fortified with Euprotin as a standard procedure.

ELIGIBILITY:
Inclusion Criteria:

* gestational age≤32 weeks and birthweight ≤1250 gr, and <48 hours postnatal age

Exclusion Criteria:

* Major congenital and/or chromosomal anomaly, Cyanotic congenital heart disease, Asphyxiated birth with pH <7.0 and base deficit ≥16mmol/l Severe cardiopulmonary compromise or multiorgan failure Twin-twin transfusion, Those died in postnatal 5 days of age

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 199 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
incidence of feeding intolerance | 28 days
  incidence of feeding intolerance
time to reach full enteral feedings sustained for 72 hours. | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak Women's Health and Education Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Bozkurt O, Alyamac Dizdar E, Bidev D, Sari FN, Uras N, Oguz SS. Prolonged minimal enteral nutrition versus early feeding advancements in preterm infants with birth weight </=1250 g: a prospective randomized trial. J Matern Fetal Neonatal Med. 2022 Jan;35(2):341-347. doi: 10.1080/14767058.2020.1716723. Epub 2020 Jan 29. PMID 31994953